CLINICAL TRIAL: NCT07212712
Title: The Role of Estrogen and Testosterone in Determining Brain Blood Flow and Metabolic Regulation in Humans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Phil Ainslie, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H25-00385
Record Dates: First submitted 2025-09-24; First posted 2025-10-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cerebral Blood Flow; Cerebral Blood Flow Regulation; Sex Differences; Exercise; Vascular
MeSH Terms: conditions — Motor Activity | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Estradiol; Testosterone; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hormone Manipulation (Experimental): Participants will act as their own controls, completing the experiment 3 times. First, with no hormone manipulation; second, with blockade of hormone production; third, with hormone add-back.
  Interventions: Drug: GnRH antagonist; Drug: Estradiol (E2); Drug: Testosterone; Drug: Anastrozole (Arimidex)

INTERVENTIONS:
Drug: GnRH antagonist — blockade of hormone production
Drug: Estradiol (E2) — Estrogen add-back in females
Drug: Testosterone — testosterone add-back in males
Drug: Anastrozole (Arimidex) — Prevention of testosterone conversion to estrogen in males

SUMMARY:
Due to historical exclusion of females from research, there are gaps in the understanding of female physiology, how it differs from males, and how sex-specific hormones contribute. As a result, many diagnoses and treatments are based on male physiology and may not be appropriate or effective for females. Females consistently experience greater risk and report worse neurological outcomes in many diseases, including stroke, cardiac arrest, and dementia. As research in females progresses, differences between sexes and changes throughout the lifespan (e.g., puberty, menopause) highlight the importance of understanding the effects of sex and sex-specific hormones on the body. The brain is arguably the most important organ in the body, consuming 20% of the body's total energy. Previous research supports higher blood flow to the brain in females, and research in animals suggests hormones such as estrogen, progesterone, and testosterone are responsible. However, it is extremely difficult to isolate these hormones in humans, due to natural fluctuations (i.e., menstrual cycle). Therefore, the investigators plan to explore the direct role of these sex-specific hormones in regulating blood flow to the brain by blocking hormone production in healthy males and females and giving back testosterone and estrogen, respectively. The investigators will then conduct a range of tests to look at blood flow to the brain at rest and during various stressors. This research will provide crucial insight into how males and females differ in regulation of brain blood flow and inform new treatments and therapies to a wide range of brain injuries and diseases, improving outcomes and reducing the sex disparity in clinical pathways.

DETAILED DESCRIPTION:
Sex hormones have been demonstrated to influence cardiovascular function in humans and cerebrovascular function in preclinical models. Declines in gonadal function have been attributed to the development of chronic disease risk in humans, including stroke, cognitive decline and dementia but the pathophysiology of these disorders remains unclear, in part, because there remains a gap-in-knowledge of the regulatory actions of sex hormones on cerebrovascular function in males and females. Therefore, the major goal of this application is to determine the independent regulatory actions of testosterone and estradiol on cerebrovascular function in males and females, respectively. Determination of this fundamental physiology is needed to inform future studies evaluating the sex-specific pathology physiology of chronic diseases and/or the development of efficacious sex-specific interventions for improving chronic disease risk.

To the investigator's knowledge, there is minimal evidence in humans isolating the influence of these hormones on basic mechanisms of brain blood flow regulation in vivo. Cross-sectional studies demonstrate younger females show significantly higher resting cerebral blood flow (CBF) compared to young males however, this sex difference in CBF is lost after midlife. This loss of female 'protection' on CBF is often attributed to hormonal differences following menopause. Further evidence in animal models support a key role of estrogen in both resting CBF and reactivity. Crucially, these findings have not been replicated in humans, due to natural fluctuations in sex hormones. Research investigating natural hormonal fluctuations throughout the menstrual cycle and menopause provides conflicting findings, falling short on isolating the specific hormonal influences on cerebrovascular physiology likely due large interindividual variations in hormone levels and cycle lengths.

Similarly, the presence of normal physiological levels of testosterone has been shown to influence chronic disease risk including cardiovascular disease risk and peripheral vascular function. However, whether testosterone concentrations influence CBF in males remains incompletely understood with one study showing testosterone may enhance CBF in older hypogonadal men. Furthermore, testosterone can be converted to estradiol via a specific enzyme, aromatase; thus, it is unclear whether the findings of prior study were related to changes in testosterone or estradiol concentrations in hypogonadal males. A definitive role of these hormones in brain blood flow regulation remains to be elucidated.

Current published studies suffer from several key limitations. First, many studies are unable to isolate the impact of hormones and their causality on cerebrovascular function in humans. The inability to replicate findings from direct hormone manipulation in animals with observational data during natural hormone cycling in humans suggests measuring females during their menstrual cycles is not adequate for understanding the direct role of these hormones. There is a very large degree of variation both between and within individuals throughout their menstrual cycles, proving difficult to relate changes in function with hormone levels. In males, very limited research exists investigating how testosterone influences cerebrovascular function. Further, this research will have direct implications for peri- and postmenopausal women, who are regularly prescribed exogenous estradiol for symptom management. Understanding the role of hormones in healthy physiology will allow direct translation to a myriad of hormonal disorders, including endometriosis, polycystic ovary syndrome, uterine fibroids, and hypogonadism. Individuals with endometriosis are commonly prescribed oral GnRH antagonist, which can be combined with estradiol for prolonged use (> 6 months). Similarly, males with hypogonadism often supplement testosterone for prolonged periods with minimal negative effects.

This study will allow for isolation of estradiol in females and testosterone in males to investigate their role on cerebrovascular regulation. In contrast with previous observational studies throughout the menstrual cycle and menopause in females and aging in males, this study will provide a controlled environment to determine causal relationships between hormones and physiology without the presence of confounding variables. This study will address the gap in literature between interventional models in animals and observational studies in healthy humans. This study will provide fundamental understandings of healthy physiology that will shape future studies to investigate the role of estradiol and testosterone in clinical populations.

The primary objective of this study is to determine how estrogen and testosterone influence cerebral blood flow and metabolism.

Primary Hypotheses:

* Cerebral blood flow and cerebral metabolic rate of oxygen consumption will be reduced in females with hormone blockade but augmented with estrogen add-back.
* Cerebral blood flow and cerebral metabolic rate of oxygen consumption will be increased in males with hormone blockade but attenuated with testosterone add-back.

To meet cerebral metabolic demands, the brain is dependent upon constant oxygen and nutrient delivery. Cerebral oxygen delivery is directly proportional to CBF and the arterial oxygen content (CaO2); it is widely known that CaO2 is lower in females, owing to the impact of anemia, hormones, and other related factors (e.g., hemoglobin, menses). To compensate, in order to maintain a stable cerebral oxygen delivery, females increase their resting CBF. Indeed, both CaO2 and hemoglobin levels are related to CBF levels. Very limited research has investigated whether cerebral metabolism differs between young males and females, with one study reporting a similar cerebral metabolic rate of oxygen (CMRO2), and another reporting higher CMRO2 in females. As cerebral metabolism is determined by CBF and the degree of oxygen extracted by the brain (oxygen extraction fraction; OEF), we must measure CMRO2 to appropriately interpret differences in CBF throughout our intervention.

Measuring CMRO₂ with the direct, invasive Fick method is the gold standard approach. By directly quantifying CBF and the arterial-venous difference in oxygen content, the Fick approach provides an absolute and internally consistent measure of brain oxygen consumption, rather than an indirect surrogate (as used with MRI, for example). This directness minimizes reliance on modeling assumptions and calibration factors that can introduce systematic bias in non-invasive techniques. As a result, Fick-based CMRO₂ measurements offer high accuracy and reproducibility; this approach is often used for validating newer imaging methods and for studies in which precise quantification of cerebral metabolism is essential. In terms of CBF, the majority of studies that of explored sex differences have typically incorporated measures of intracranial velocity via transcranial Doppler (TCD) rather than assessment flow. In this study, we will employ contemporary measures of Duplex ultrasound which measures extracranial flow and further validates our inclusion of CMRO2 measures.

Despite its invasiveness, the Fick method offers unique benefits that justify its use in select experimental and clinical contexts. Because it yields absolute metabolic values, the direct Fick method facilitates meaningful comparisons across subjects, conditions, and studies for the critical benchmark and gold-standard for understanding cerebral energetics. Compared with MRI-based approaches, the Fick technique quantifies CMRO2 from measured cerebral blood flow and the arterial-venous oxygen content difference, yielding an absolute metabolic rate with minimal dependence on modeling assumptions. In contrast, MRI-derived CMRO2 estimates typically rely on indirect contrasts (e.g., BOLD, ASL) and biophysical models that require assumptions about vascular geometry, baseline physiology (eg., hemoglobin levels), and coupling between flow, volume, and metabolism, all of which can vary across subjects and conditions. As a result, the invasive Fick method offers superior accuracy and interpretability, particularly when precise quantification is required or when validating MRI-based metabolic measurements. While PET imaging would be considered the gold standard to measure regional blood flow and oxygen or glucose metabolism by tracking the uptake of injected radioactive tracers (usually H₂¹⁵O), it is also invasive, requiring injected radioactive tracers and does not provide information on global CMRO2 or lactate metabolism. For a more extensive review of the limitations of PET imaging for global cerebral metabolism, please see Duffy et al. Therefore, neither PET nor MRI imaging can be easily used when common stressors are implemented (e.g., exercise, changes in partial pressures of oxygen and carbon dioxide) to provide an index of brain resilience.

ELIGIBILITY:
Inclusion Criteria:

The investigators will recruit healthy young (18-40 years) males (n = 25) and females (n = 25). Females must be naturally cycling (i.e., no oral or hormonal contraceptives), not pregnant, and premenopausal. Participants must be normotensive (<140/90 mmHg & >90/60 mmHg) and have no medical history of cerebrovascular, cardiopulmonary, cardiovascular, neuromuscular, and renal disease assessed by a study questionnaire. A recent physical examination (within 1 year of participation) from a family physician or a completed physical examination by the study doctor is required prior to participation. All subjects will sign an informed consent form prior to participation.

Participants will be excluded if they meet any of the following criteria:

* Hypertensive (≥140/90 mmHg) or hypotensive (≤90/60 mmHg)
* BMI ≥ 30 kg/m2
* Fasting blood glucose ≥ 100 mg/dL
* Abnormal results on standard blood hematology tests (e.g., complete blood count, comprehensive metabolic panel)
* Males with hypogonadism (total testosterone ≤ 262 ng/dL, per Endocrine Society recommendations)
* Any history of cerebrovascular, cardiopulmonary, cardiovascular, neuromuscular, or renal disease
* Any liver dysfunction or disease
* Taking any cardiovascular medications or medications that would interfere with study medications (e.g., strong organic anion transporting polypeptide 1B1 inhibitors)
* Contraindications or sensitivities to study medications
* Current eating disorder (defined as >2 on the 'SCOFF' questionnaire 67)
* Current smokers
* Females with an irregular menstrual cycle or any medical conditions affecting the menstrual cycle (normal cycle defined as 21-35 days from menstrual cycle diary)
* Females who are pregnant (assessed with pregnancy test at screening and prior to starting medications), breastfeeding, or planning to conceive within 3 months
* Females using hormonal birth control (Copper intrauterine devices [IUDs] will be allowed as they do not change systemic hormone levels)
* Females who are peri- or postmenopausal (as determined by STRAW criteria 68)
* History of hormone-sensitive cancers (i.e., breast, ovarian, uterine or prostate)
* Z-score < -2 as assessed with DXA scan (to determine risk of decrease in bone mineral density)
* Assessed using the Center for Epidemiologic Studies Depression (CES-D) scale, participants with a score > 16 at screening unless otherwise approved by the study MD

Ages: 18 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow responses to estrogen and testosterone | 7 days
  To determine how cerebral blood flow regulation is altered by estrogen and testosterone concentrations. Measured through doppler ultrasonography, and reported in mL/min.
Cerebral metabolic changes with estrogen and testosterone | 4 days
  Measured as cerebral metabolic rate of oxygen consumption. Determined using arterial and internal jugular vein blood sampling coupled with doppler ultrasound, to determine metabolism directly using the Fick method.

SECONDARY OUTCOMES:
Hormone influences on appetite sensations | 7 days
  How estrogen and testosterone influence appetite sensations (visual analog scale)
How estrogen and testosterone influence energy intake | 7 days
  dietary intake, measured with self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ainslie, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia - Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will share individual data from published results on request.

REFERENCES:
- [Background] Muer JD, Didier KD, Wannebo BM, Sanchez S, Khademi Motlagh H, Haley TL, Carter KJ, Banks NF, Eldridge MW, Serlin RC, Wieben O, Schrage WG. Sex differences in gray matter, white matter, and regional brain perfusion in young, healthy adults. Am J Physiol Heart Circ Physiol. 2024 Oct 1;327(4):H847-H858. doi: 10.1152/ajpheart.00341.2024. Epub 2024 Aug 9. PMID 39120466
- [Background] Reeves MJ, Bushnell CD, Howard G, Gargano JW, Duncan PW, Lynch G, Khatiwoda A, Lisabeth L. Sex differences in stroke: epidemiology, clinical presentation, medical care, and outcomes. Lancet Neurol. 2008 Oct;7(10):915-26. doi: 10.1016/S1474-4422(08)70193-5. Epub 2008 Aug 21. PMID 18722812
- [Background] Moreau KL, Hildreth KL, Klawitter J, Blatchford P, Kohrt WM. Decline in endothelial function across the menopause transition in healthy women is related to decreased estradiol and increased oxidative stress. Geroscience. 2020 Dec;42(6):1699-1714. doi: 10.1007/s11357-020-00236-7. Epub 2020 Aug 8. PMID 32770384